CLINICAL TRIAL: NCT03569345
Title: Investigation of Local Skin Reactions and Safety After Combined Treatment of Basal Cell Carcinoma Using Ablative Fractional Laser and Ingenol Mebutate - an Exploratory, Prospective, Open-label Phase 2a Trial.
Brief Title: Basal Cell Carcinomas Treated With Ablative Fractional Laser and Ingenol Mebutate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merete Haedersdal (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, Professor, Senior Consultant, PhD, DMSc, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT-nr: 2017-002843-14
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm (Experimental): Basal cell carcinoma (BCC) patients Patients (>18 pr) with histologically-verified superficial or nodular basal cell carcinoma (<20 mm on face/scalp, <50 mm on trunk/extremities)
  Interventions: Drug: AFXl-assisted ingenol mebutate delivery

INTERVENTIONS:
Drug: AFXl-assisted ingenol mebutate delivery — Patients will receive ablative fractional laser (AFXl)-assisted ingenol mebutate (IM) as a treatment for their cutaneous basal cell carcinoma (BCC). Treatment areas consisting of tumors and a 5 mm margin will undergo AFXl exposure (CO2 laser) followed by IM 0.015% or 0.05% under occlusion for 2-3 days. .
  local skin reactions are monitored at baseline (day1), day 3/4, day 8, day 15, day 29, day 90, and tumor response monitored at baseline, day 29, and day 90. An additional repeat AFXl-IM treatment on day 29 will be offered if tumors persist, based on clinical evaluation and imaging on day 30.

SUMMARY:
A prospective clinical, uncontrolled, open-label, explorative phase 2a trial on patients with histologically-confirmed superficial and nodular basal cell carcinoma (BCC). The study assesses tolerability and tumor clearance after laser-assisted topical delivery of topical ingenol mebutate.

DETAILED DESCRIPTION:
Patients will receive ablative fractional laser (AFXl)-assisted ingenol mebutate (IM) as a treatment for their cutaneous basal cell carcinoma (BCC). Treatment areas consisting of tumors and a 5 mm margin will undergo AFXl exposure (CO2 laser) followed by IM 0.015% or 0.05% under occlusion for 2-3 days. .

local skin reactions are monitored at baseline (day1), day 3/4, day 8, day 15, day 29, day 90, and tumor response monitored at baseline, day 29, and day 90. An additional repeat AFXl-IM treatment on day 29 will be offered if tumors persist, based on clinical evaluation and imaging on day 30.

Primary outcome:

1. severity and duration of clinical local skin reactions including erythema, scaling, edema, blistering, erosion/ulceration and crusting using a 0-4-point scale at all visits from baseline to day 90.
2. To monitor BCC tumor response on clinical assessments supported by non-invasive imaging techniques including optical coherence tomography (OCT) and reflectance confocal microscopy (RCM) at baseline, day 29 and day 90.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are eligible to participate in this study

* Patients with histologically verified, low-risk, previously untreated superficial or nodular BCCs on the scalp, face, extremities or trunk
* > 18 years of age at baseline
* Legally competent, able to give verbal and written consent
* Communicate in Danish verbally as well as in writing
* Subject in good general health, is willing to participate and able to give informed consent, and can comply with protocol requirements.
* Fitzpatrick skin phototype I-III
* Female subjects of childbearing potential must be confirmed not pregnant by a negative urine pregnancy test prior to trial treatment.

Exclusion Criteria:

Subjects meeting any one of the following criteria are not eligible to participate in this study

* Patients with

  o High-risk BCC
* Tumors on the following anatomical locations:

  * Midface region
  * Orbital areas
  * Ears
* ii. Size:
* > 20 mm in facial/scalp areas
* > 50 mm in non-facial/non-scalp areas

  * Subtype:
  * Morpheaform
  * Medical history
* Gorlin syndrome

  o Immunosuppressive medication
* Subjects with a known allergy to IM.
* Individuals with other skin diseases in the area of research interest
* Subjects with tattoo in the treatment area which may interfere with or confound evaluation of the study
* Subjects with a history of keloids which is deemed clinically relevant in the opinion of the investigator
* Subjects with Fitzpatrick skin phototype IV-VI
* Lactating or pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Change in occurrence of local skin reactions | 0-90 days
  Non-blinded, clinical evaluation of local erythema, edema, flaking, crusting/scabbing, pustulation, scarring, hypo(hyperpigmentation, infection in treated areas will be performed by physician using an FDA-approved 0-4 point lsr scale at day 1, 3/4, 8, 15, 29 and 90 after AFXl exposure. Standardized, clinical photographs are taken to document skin reactions at each visit

SECONDARY OUTCOMES:
Tumor response clinically | baseline, day 29, day 90
  Tumor clearance (yes or no) will be evaluated clinically at baseline, at day 29 and day 90. If residual tumor is identified at day 90 patients will receive conventional treatment according to national guidelines.
Tumor response by imaging techniques | baseline, day 29, day 90
  Clearance (yes or no) will be evaluated using non-invasive reflectance confocal microscopy and optical coherence tomography at baseline, day 30 and day 90.f residual tumor is identified at day 90 patients will receive conventional treatment according to national guidelines.
Tumor response - histology | At day 90
  HIstological verification of tumor clearance will be performed at day 90 after first treatment using tissue sections from a punch biopsy (up to 4 mm). If residual tumor is identified at day 90 patients will receive conventional treatment according to national guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermtology, Bispebjerg University Hospital, Copenhagen, Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided